CLINICAL TRIAL: NCT05671380
Title: A Pragmatic Trial of Chronic Disease Approaches to Ameliorate Tobacco Related Cardiovascular Disease Health Disparities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00013870
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use Cessation; Cardiovascular Diseases; Tobacco Use; Smoking; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Cessation; Cardiovascular Diseases; Tobacco Use; Smoking; Smoking Cessation | interventions — Lactoperoxidase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care: Ask-Advice-Connect (AAC) (Active Comparator): AAC participants will receive care through their primary care provider as usual (with the caveat that providers in the clinics will be trained to provide AAC). AAC includes enhanced access to State Quitline and Nicotine Replacement Therapy.
  Interventions: Behavioral: Ask-Advice-Connect (AAC)
- AAC + Longitudinal Proactive Outreach (LPO) (Experimental): AAC+LPO participants will receive AAC plus an MI tailored outreach call at baseline and at 3, 6, and 9 months post-enrollment. AAC includes enhanced access to State Quitline and Nicotine Replacement Therapy.
  Interventions: Behavioral: Longitudinal Proactive Outreach (LPO).; Behavioral: Ask-Advice-Connect (AAC)

INTERVENTIONS:
Behavioral: Longitudinal Proactive Outreach (LPO). — All participants will receive personalized invitation materials (in their preferred language) with messages culturally and linguistically tailored to BIPOC communities, guided by the literature on culturally adapting evidence-based interventions. The study team will tailor these resources in collaboration with the CE core. The tailored mailed packet will include an invitation letter and a brochure describing the types of tobacco treatment services available from their health system and from Quit Partner. One week after the written materials are sent, participants assigned to this condition will receive LPO by a MI-trained coach. The MI outreach call protocol will consist of 6 contact attempts over two weeks.The MI outreach call protocol will be repeated at 3, 6, and 9 months for a total of four outreach cycles because participants may not have quit or may have relapsed.
  Arms: AAC + Longitudinal Proactive Outreach (LPO)
Behavioral: Ask-Advice-Connect (AAC) — Licensed Practical Nurses will be trained to ask all patients if they smoke, document smoking status in the EHR, advise patients to stop smoking, and complete an electronic referral to Quit Partner or the smoking cessation clinic. AAC will be designed to connect participants to Quit Partner Minnesota to receive tobacco cessation counseling. Quit Partner™ is a family of programs available to help Minnesota residents quit commercial tobacco, administered by the Minnesota Department of Health (MDH). Quit Partner programs are provided by National Jewish Health (NJH). Any Minnesota resident can access a free 2-week supply of Nicotine Replacement Therapy (NRT). Uninsured and underinsured residents can access the full Quit Partner programs, including free one-on- one coaching, more NRT, and additional supports. Quit Partner also offers four population- specific programs and calls are available in several languages.

SUMMARY:
This project will evaluate a proactive outreach intervention for tobacco cessation among primary care BIPOC populations who smoke in two health systems across the region. Compared with Whites, BIPOC populations in the US experience disproportionate health consequences from commercial cigarette use. Few evidence-based cessation treatments (EBCTs) have been specifically developed, evaluated, or implemented for BIPOC populations. Moreover, uptake of EBCT (e.g. medication, counseling) is lower among BIPOC populations. Reasons for the failure to engage BIPOC patients in EBCTs are complex and multi-level (e.g., patient, provider, healthcare system). To address these gaps, the investigators will assess the added effectiveness of an approach to augment the standard of care with longitudinal proactive outreach to connect BIPOC adults with EBCT. The proposed multi-level intervention leverages the electronic health record to identify patients who smoke, who can then be proactively engaged via culturally tailored outreach to connect them to EBCT. The proactive approach may circumvent experiences of bias within the healthcare system and thus enhance engagement.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking BIPOC patients within the Hennepin Healthcare or MCHS system. BIPOC patients are any patients with a chart identified race that is not White, and will be verified by self-report from the baseline survey.
* Currently smoke >1 cigarette over the past 30 days
* Must have address or telephone number in the electronic health record

Exclusion Criteria:

* Electronic health record documented cognitive impairment or legal guardianship
* Patients who have opted out of reserach studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
7-day point-prevalence smoking abstinence at 18 months | 18 months
  7-day point prevalence abstinence from combustible tobacco will be verified at 18 months post-enrollment. Surveys to self-report abstinence will be provided at 6, 12, and 18 months.
  Self-reported smoking abstinence will be verified using expired carbon monoxide as the primary method with salivary cotinine as an alternative method at the 18-month follow-up. Participants with a CO of < 6 ppm will be considered abstinent. Participants with a salivary cotinine < 10 ng/ml will be considered abstinent.

SECONDARY OUTCOMES:
Change in Theory of Planned Behavior Questionnaire (TPB-Q) Score | 0, 6, 12, and 18 months
  The TPB-Q is a commonly used and thoroughly validated instrument that maps onto the three predictors of health behavior change in the Theory of Planned Behavior: attitudes about the behavior, perceived subjective norms about the behavior, and perceived control over the behavior. The TPB-Q items have common wording tapping into those three domains, but the scale was developed such that the items are customized to the specific behavioral goal of an intervention, and thus still comparable across behaviors.
Change in Treatment utilization. | 6, 12, and 18 months
  Self-reported utilization of evidence-based cessation treatment (EBCT) will be assessed during the 18-month follow-up from any source. The main treatment outcome will be initiation of counseling with Quit Partner or the participant's healthcare provider, combined with medication treatment utilization. Initiation of counseling treatment with the Quit Partner will be defined as completion of a warm transfer or electronic referral to the quitline. Initiation of medication treatment will be defined as using one or more tobacco dependence medications (e.g., NRT, bupropion or varenicline) in the 18-month follow-up period. Additional treatment utilization outcomes include individual use of counseling or medication and use of any form of EBCT.
Change in Overall Quality of Life | 0, 6, 12, and 18 months
  Overall quality of life will be assessed using a single-item numerical linear analogue self-assessment from 0 (as bad as it can be) to 10 (as good as it can be) via survey through 18 months post-enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fu, MD, MSCE, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (3):
- United States (3):
  - Hennepin Healthcare, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Health System, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu SS, Hammett P, Nelson D, Busch A, McKinney W, Sharma P, Patten CA, Gutierrez Sacasa N, Andreae L, Japuntich S. Evaluating chronic disease approaches to ameliorate tobacco-related health disparities: Study protocol of a hybrid type 1 implementation-effectiveness trial. Contemp Clin Trials Commun. 2024 Oct 16;42:101380. doi: 10.1016/j.conctc.2024.101380. eCollection 2024 Dec. PMID 39498443